CLINICAL TRIAL: NCT02409251
Title: Requesting Behaviour of Rheumatologists Regarding Antinuclear Antibodies (ANA) in Patients With Rheumatologic Complaints
Brief Title: Rheumatologists and the Requesting of Antinuclear Antibodies (ANA) Tests in Patients With Rheumatologic Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Principal Investigator, Nienke Lesuis, MD, Sint Maartenskliniek
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RR-103-ANA
Record Dates: First submitted 2015-03-09; First posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatic Diseases
Keywords: Antinuclear antibody (ANA); Overuse; Rheumatologists; Quality of care
MeSH Terms: conditions — Rheumatic Diseases | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education and feedback (Experimental): The intervention consisted of a one-hour, small group educational session. During this session information on rational ANA testing was provided and feedback on current ANA testing was provided to the rheumatologists. A booster session with the same components was held 6 months after the first session.
  Interventions: Behavioral: Education and feedback

INTERVENTIONS:
Behavioral: Education and feedback

SUMMARY:
The aim of this study is to assess the effect of a simple intervention (a combination of education and feedback) on Antinuclear Antibody (ANA) testing.

This aim was chosen because of the known overuse of many laboratory tests, of which ANA testing is one. As overuse of ANA tests can have negative consequences (both for patients and society), the investigators designed an intervention to see how this would influence Antinuclear Antibody testing by rheumatologists.

ELIGIBILITY:
Inclusion Criteria rheumatologists:

* rheumatologists who are consulting patients at the rheumatology outpatient clinic of a participating centre

Exclusion Criteria rheumatologists:

* rheumatologists not working the full study period (pre- and post-intervention) at a participating centre
* rheumatologists not giving their consent to participate

Inclusion Criteria patients - all patients with an ANA test requested by an included rheumatologist during the study period

Exclusion Criteria patients

- patients with an ANA test requested during a clinical admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline (pre-intervention) ANA/new patient ratio (APR) at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Number of ANA tests divided by the number of new patients
Change from baseline (pre-intervention) % of positive ANA tests at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Percentage of ANA tests reported as positive by the local laboratory. ANA tests reported as 'weakly positive' are regarded as negative.
Change from baseline (pre-intervention) % of repeated ANA testing at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Percentage of patients with ≥1 ANA test in 12 months (pre- or post-intervention period)
Change from baseline (pre-intervention) % of ANA associated diagnoses at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Percentage of patients, in which an ANA is done during the study period, with final diagnosis of SLE, SSc, PM/DM, MCTD or SS
Change from baseline (pre-intervention) APR variation between rheumatologists at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Standard deviation around the mean APR, calculated from the APRs of the individual rheumatologists
Change from baseline (pre-intervention) reaching the of target APR at 12 months (post-intervention) | Pre- and post-intervention (both 12 months)
  Difference (percentage) between the actual APR and the target-APR defined during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ronald van Vollenhoven, MD, PhD, Principal Investigator — Karolinska Institutet; Marlies Hulscher, PhD, Principal Investigator — Scientific Institute for Quality of Healthcare, Radboud University Medical Center, Nijmegen, the Netherlands; Alfons den Broeder, MD, PhD, Principal Investigator — Sint Maartenskliniek, Nijmegen, the Netherlands
Locations (3):
- Netherlands (3):
  - Sint Maartenskliniek, Nijmegen, Gelderland
  - Radboud University Medical Center, Nijmegen
  - Maartenskliniek Woerden, Woerden

REFERENCES:
- [Derived] Lesuis N, Hulscher ME, Piek E, Demirel H, van der Laan-Baalbergen N, Meek I, van Vollenhoven RF, den Broeder AA. Choosing Wisely in Daily Practice: An Intervention Study on Antinuclear Antibody Testing by Rheumatologists. Arthritis Care Res (Hoboken). 2016 Apr;68(4):562-9. doi: 10.1002/acr.22725. PMID 26414008